CLINICAL TRIAL: NCT00003467
Title: Phase II Treatment of Adults With Recurrent Supratentorial Low Grade Glioma With Gliadel Wafers
Brief Title: Carmustine in Treating Adults With Recurrent Supratentorial Low-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Henry Friedman, MD, Duke UMC
Purpose: Treatment
Other Study IDs: 1706; DUMC-1706-02-9R5; DUMC-1706-01-9R4; DUMC-000693-00-4; DUMC-1509-97-10; DUMC-1568-98-10R1; DUMC-1706-00-9R3; DUMC-97131; NCI-G98-1470; CDR0000066503 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult brain stem glioma; adult mixed glioma; adult anaplastic astrocytoma; adult pilocytic astrocytoma; adult oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioma; Astrocytoma; Oligodendroglioma | interventions — Carmustine; Surgical Procedures, Operative

INTERVENTIONS:
Drug: carmustine
Drug: polifeprosan 20 with carmustine implant
Procedure: surgical procedure

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of carmustine in treating adults with recurrent supratentorial low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of Gliadel wafers (carmustine) in the treatment of recurrent supratentorial low grade glioma.
* Assess the toxicity of this therapy in these patients.

OUTLINE: Patients are stratified by disease (fibrillary astrocytoma vs oligodendroglioma or mixed glioma).

Patients receive up to 8 Gliadel wafers (containing carmustine) implanted in the resected tumor cavity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: This study will accrue a maximum of 68 patients within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent primary low grade glioma including:

  * Fibrillary astrocytoma
  * Oligodendroglioma
  * Mixed glioma
* Evidence of measurable enhancing or non-enhancing CNS neoplasm on MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Hematocrit greater than 29%
* Absolute neutrophil count greater than 1500/mm^3
* Platelet count greater than 125,000/mm^3

Hepatic:

* SGOT less than 1.5 times upper limit of normal (ULN)
* Bilirubin less than 1.5 times ULN

Renal:

* Creatinine less than 1.5 mg/dL
* BUN less than 25 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy unless disease progression

Endocrine therapy:

* Concurrent corticosteroids allowed (must be on stable dose for 1 week prior to study)
* No concurrent immunosuppressive agents

Radiotherapy:

* At least 4 weeks since prior radiotherapy unless disease progression

Surgery:

* Not specified

Other:

* No other concurrent medication that may interfere with study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 1998-01; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States